CLINICAL TRIAL: NCT02317588
Title: Gender Effects of Dietary Omega-3 Fatty Acids From Plant and Marine Sources on Oxylipins in Healthy Humans
Acronym: OXGEN-2014
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Manitoba Health Research Council (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B2014:036
Record Dates: First submitted 2014-12-11; First posted 2014-12-16 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Healthy
Keywords: Oxylipins; Flax oil; Fish oil
MeSH Terms: interventions — Linseed Oil; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flax Oil (Active Comparator): Flax oil 4 grams of ALA per day for 28 days (4 weeks).
  Interventions: Dietary Supplement: Flax Oil
- Fish Oil (Active Comparator): Fish oil at a dose of 4 grams DHA + 0.8 grams EPA per day for 28 days (4 weeks).
  Interventions: Dietary Supplement: Fish Oil

INTERVENTIONS:
Dietary Supplement: Flax Oil — Participants will consume capsules containing flax oil at a dose of 4 grams of ALA per day (8 capsules a day) with a meal for 28 days (4 weeks).
  Other Names: Now Brand Organic Flax Oil
  Arms: Flax Oil
Dietary Supplement: Fish Oil — Participants will consume capsules containing fish oil at a dose of 4 grams DHA + 0.8 grams EPA per day (8 capsules) for 28 days (4 weeks).
  Other Names: Carlson DHA Gems
  Arms: Fish Oil

SUMMARY:
This study is single site, double-blind, randomized, cross-over study designed to compare the effects of flax oil and fish oil supplementation on the oxylipin profile in healthy males and females. Eligible participants will complete two (2) Supplementation Phases (flax oil versus fish oil) and will be asked to attend 6 in-person clinic visits (0, 1, 3, 7, 14 and 28 days) for blood and urine collection during each phase. Participants will consume 8 capsules a day for 28 days containing either A) Flax Oil at 4 grams of ALA per day ,in one phase and B) Fish Oil at a dose of 4 grams DHA + 0.8 grams EPA per day in the next phase. Participants will be randomized and blinded and will therefore no know what supplement they are taking in either phase.

DETAILED DESCRIPTION:
This is a single site, double-blind, randomized, crossover study designed to compare the effects of dietary omega-3 fatty acids from flax oil versus fish oil supplementation on oxylipin profiles over time (0 to 4 weeks) and between healthy males and females.

Recruitment will consist of a total of six (6) male and six (6) female participants. Participants will be recruited through advertisement from the local community. The study will be conducted at the Asper Centre for Clinical Research, St. Boniface Hospital. Participants will be asked to provide written informed consent prior to participation in the study. Participants who have provided written consent will be asked to attend an in-patient visit to provide a fasting blood sample. Should the participant be eligible to participate, they will be scheduled for a minimum 6 week Run-in Period, a 4 week Supplementation Phase, a minimum 6 week Wash-out Period and then a second 4 week Supplementation Phase; each Supplementation Phase will have 6 in-person visits (0, 1, 3, 7, 14 and 28 days) to obtain fasting blood and urine samples and for completion of the Study Checklist. During each 4 week Supplementation Phase, participants will consume capsules containing flax oil and at a dose of 4 grams of ALA/day, or capsules containing fish oil and at a dose of 4 grams DHA + 0.8 grams EPA/day. A 3-Day Food Record and Activity Questionnaire will be completed before the Day 0 visit and during week 3 of each Supplementation Phase.

Provision of flax oil or fish oil in capsules will allow this study to be double-blinded. Blinding will reduce potential bias during data collection and evaluation of study endpoints. Both the research team and the participant are blinded from the time of randomization and for the duration of the study. Randomization will be used to avoid bias in the assignment; to increase the likelihood that known and unknown participant characteristics are evenly balanced across the various test groups; and to enhance the validity of statistical comparisons across test groups.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet the following criteria to be eligible for participation in the study:

1. Male, or non-pregnant, non-lactating premenopausal female, ≥18 and ≤50 years of age;
2. Normal blood lipid profile (total cholesterol <5.2 mmol/L, LDL-cholesterol <3.4 mmol/L, HDL-cholesterol >0.9 mmol/L, triglycerides <1.7 mmol/L), plasma creatinine <1.5× upper limit of normal (ULN) where the normal range is 50-97 µmol/L, and glycated hemoglobin <6%; aspartate transaminase (AST) <2× ULN where the normal range is 10 - 32 U/L, and alanine transaminase (ALT) <2× ULN where the normal range is <25 U/L;
3. Blood pressure <140/90;
4. Body mass index (BMI) of 18 to 28;
5. Stable regime if taking vitamin and mineral/dietary/herbal supplements for the past 1 months and while participating in the study;
6. Willing to maintain a stable level of activity while participating in the study;
7. Willing to maintain dietary routine and to refrain from consuming omega-3 supplements or omega-3 rich foods (>0.3 grams ALA/serving, or >0.1 grams EPA + DHA/serving) from acceptance into the study until the final study visit;
8. Females must have normal menses and can be on birth control;
9. Agrees to not donate blood while participating in the study and for 2 months after participation in the study.
10. Willing to comply with the protocol requirements and procedures;
11. Willing to provide informed consent.

Exclusion Criteria:

Participants will be excluded if they have any of the following:

1. Presence of a clinically diagnosed disease affecting the circulatory, respiratory, immune, skeletal, urinary, muscular, endocrine, digestive, nervous or reproductive system, or a disease condition that has required or currently requires medical treatment;
2. Taking any prescribed medication, regular use of acetylsalicylic acid (e.g. Aspirin), ibuprofen (e.g. Advil) or acetaminophen (e.g. Tylenol) within the last 3 months;
3. Allergy or sensitivity to any of the study product ingredients, such as flax, flax oil, or marine source oils such as fish or shellfish.
4. Cigarette/cigar smoking or use of tobacco products within the past 12 months or during the study;
5. Body weight has not been stable (±3 kg) over the past 6 months;
6. Consumption of >15 alcoholic beverages per week (according to Canada's Low-Risk Alcohol Drinking Guidelines, 2012) within the last 3 months or while participating in the study;
7. Current (within the past 30 days) bacterial, viral or fungal infection;
8. Unable to obtain blood sample at the screening and/or week 0 visit.
9. Donated or had blood collected in the 2 months prior to participation the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Plasma oxylipin concentrations over time | 28 Days
  A fasting venous blood sample will be obtained from the participant on Days 0, 1, 3, 7, 14 and 28 of each 'Supplementation Phase' for the assessment of plasma oxylipin profile.

SECONDARY OUTCOMES:
Fatty Acid Composition Over Time | 28 Days
  A fasting venous blood sample will be obtained from the participant on Days 0, 1, 3, 7, 14 and 28 of each 'Supplementation Phase' for the assessment of fatty acid composition.
Assessment of Markers of Metabolism, Oxidative Stress & Inflammation Over Time | 28 Days
  A fasting venous blood sample will be obtained from the participant at Day 0, 1, 3, 7, 14 and 28 of each Supplementation Phase for assessment of markers of markers of metabolism, oxidative stress and inflammation.

OTHER OUTCOMES:
Assessment of Blood Lipids Day 0 vs. Day 28 | 28 Days
  At the Day 0 and 28 visits, additional blood fasting venous blood will be obtained from the participant for measurement of total cholesterol, LDL-cholesterol, HDL-cholesterol, and triglycerides.
Comparison of Serum Oxylipins vs. Plasma Oxylipins | 28 Days
  At the Day 0 and 28 visits a fasting venous blood will be obtained for comparison of oxylipins in clotted (serum) versus unclotted (plasma) samples.

CONTACTS AND LOCATIONS:
Overall Officials: Carla Taylor, PhD, Principal Investigator — University of Manitoba
Locations (1):
- St. Boniface General Hospital, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Kakutani S, Kawashima H, Tanaka T, Shiraishi-Tateishi A, Kiso Y. Uptake of dihomo-gamma-linolenic acid by murine macrophages increases series-1 prostaglandin release following lipopolysaccharide treatment. Prostaglandins Leukot Essent Fatty Acids. 2010 Jul;83(1):23-9. doi: 10.1016/j.plefa.2010.02.032. Epub 2010 Mar 26. PMID 20347284
- [Background] Wang X, Lin H, Gu Y. Multiple roles of dihomo-gamma-linolenic acid against proliferation diseases. Lipids Health Dis. 2012 Feb 14;11:25. doi: 10.1186/1476-511X-11-25. PMID 22333072
- [Background] Harkewicz R, Fahy E, Andreyev A, Dennis EA. Arachidonate-derived dihomoprostaglandin production observed in endotoxin-stimulated macrophage-like cells. J Biol Chem. 2007 Feb 2;282(5):2899-910. doi: 10.1074/jbc.M610067200. Epub 2006 Nov 29. PMID 17135246
- [Background] Levy BD. Resolvins and protectins: natural pharmacophores for resolution biology. Prostaglandins Leukot Essent Fatty Acids. 2010 Apr-Jun;82(4-6):327-32. doi: 10.1016/j.plefa.2010.02.003. Epub 2010 Mar 15. PMID 20227865
- [Background] Serhan CN, Chiang N, Van Dyke TE. Resolving inflammation: dual anti-inflammatory and pro-resolution lipid mediators. Nat Rev Immunol. 2008 May;8(5):349-61. doi: 10.1038/nri2294. PMID 18437155
- [Background] Quehenberger O, Armando AM, Brown AH, Milne SB, Myers DS, Merrill AH, Bandyopadhyay S, Jones KN, Kelly S, Shaner RL, Sullards CM, Wang E, Murphy RC, Barkley RM, Leiker TJ, Raetz CR, Guan Z, Laird GM, Six DA, Russell DW, McDonald JG, Subramaniam S, Fahy E, Dennis EA. Lipidomics reveals a remarkable diversity of lipids in human plasma. J Lipid Res. 2010 Nov;51(11):3299-305. doi: 10.1194/jlr.M009449. Epub 2010 Jul 29. PMID 20671299
- [Background] Psychogios N, Hau DD, Peng J, Guo AC, Mandal R, Bouatra S, Sinelnikov I, Krishnamurthy R, Eisner R, Gautam B, Young N, Xia J, Knox C, Dong E, Huang P, Hollander Z, Pedersen TL, Smith SR, Bamforth F, Greiner R, McManus B, Newman JW, Goodfriend T, Wishart DS. The human serum metabolome. PLoS One. 2011 Feb 16;6(2):e16957. doi: 10.1371/journal.pone.0016957. PMID 21359215
- [Background] Schuchardt JP, Schmidt S, Kressel G, Dong H, Willenberg I, Hammock BD, Hahn A, Schebb NH. Comparison of free serum oxylipin concentrations in hyper- vs. normolipidemic men. Prostaglandins Leukot Essent Fatty Acids. 2013 Jul;89(1):19-29. doi: 10.1016/j.plefa.2013.04.001. Epub 2013 May 19. PMID 23694766
- [Background] Ramsden CE, Ringel A, Feldstein AE, Taha AY, MacIntosh BA, Hibbeln JR, Majchrzak-Hong SF, Faurot KR, Rapoport SI, Cheon Y, Chung YM, Berk M, Mann JD. Lowering dietary linoleic acid reduces bioactive oxidized linoleic acid metabolites in humans. Prostaglandins Leukot Essent Fatty Acids. 2012 Oct-Nov;87(4-5):135-41. doi: 10.1016/j.plefa.2012.08.004. Epub 2012 Sep 5. PMID 22959954
- [Background] Caligiuri SP, Love K, Winter T, Gauthier J, Taylor CG, Blydt-Hansen T, Zahradka P, Aukema HM. Dietary linoleic acid and alpha-linolenic acid differentially affect renal oxylipins and phospholipid fatty acids in diet-induced obese rats. J Nutr. 2013 Sep;143(9):1421-31. doi: 10.3945/jn.113.177360. Epub 2013 Jul 31. PMID 23902961
- [Background] Keenan AH, Pedersen TL, Fillaus K, Larson MK, Shearer GC, Newman JW. Basal omega-3 fatty acid status affects fatty acid and oxylipin responses to high-dose n3-HUFA in healthy volunteers. J Lipid Res. 2012 Aug;53(8):1662-9. doi: 10.1194/jlr.P025577. Epub 2012 May 24. PMID 22628615
- [Background] Harris WS, Mozaffarian D, Rimm E, Kris-Etherton P, Rudel LL, Appel LJ, Engler MM, Engler MB, Sacks F. Omega-6 fatty acids and risk for cardiovascular disease: a science advisory from the American Heart Association Nutrition Subcommittee of the Council on Nutrition, Physical Activity, and Metabolism; Council on Cardiovascular Nursing; and Council on Epidemiology and Prevention. Circulation. 2009 Feb 17;119(6):902-7. doi: 10.1161/CIRCULATIONAHA.108.191627. Epub 2009 Jan 26. No abstract available. PMID 19171857
- [Background] Czernichow S, Thomas D, Bruckert E. n-6 Fatty acids and cardiovascular health: a review of the evidence for dietary intake recommendations. Br J Nutr. 2010 Sep;104(6):788-96. doi: 10.1017/S0007114510002096. Epub 2010 Jun 4. PMID 20522273
- [Background] Khaw KT, Friesen MD, Riboli E, Luben R, Wareham N. Plasma phospholipid fatty acid concentration and incident coronary heart disease in men and women: the EPIC-Norfolk prospective study. PLoS Med. 2012;9(7):e1001255. doi: 10.1371/journal.pmed.1001255. Epub 2012 Jul 3. PMID 22802735
- [Background] MacLean CH, Mojica WA, Morton SC, Pencharz J, Hasenfeld Garland R, Tu W, Newberry SJ, Jungvig LK, Grossman J, Khanna P, Rhodes S, Shekelle P. Effects of omega-3 fatty acids on lipids and glycemic control in type II diabetes and the metabolic syndrome and on inflammatory bowel disease, rheumatoid arthritis, renal disease, systemic lupus erythematosus, and osteoporosis. Evid Rep Technol Assess (Summ). 2004 Mar;(89):1-4. No abstract available. PMID 15133890
- [Background] Miles EA, Calder PC. Influence of marine n-3 polyunsaturated fatty acids on immune function and a systematic review of their effects on clinical outcomes in rheumatoid arthritis. Br J Nutr. 2012 Jun;107 Suppl 2:S171-84. doi: 10.1017/S0007114512001560. PMID 22591891
- [Background] Goldberg RJ, Katz J. A meta-analysis of the analgesic effects of omega-3 polyunsaturated fatty acid supplementation for inflammatory joint pain. Pain. 2007 May;129(1-2):210-23. doi: 10.1016/j.pain.2007.01.020. Epub 2007 Mar 1. PMID 17335973
- [Background] Robinson LE, Buchholz AC, Mazurak VC. Inflammation, obesity, and fatty acid metabolism: influence of n-3 polyunsaturated fatty acids on factors contributing to metabolic syndrome. Appl Physiol Nutr Metab. 2007 Dec;32(6):1008-24. doi: 10.1139/H07-087. PMID 18059573
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Marcantoni E, Di Francesco L, Totani L, Piccoli A, Evangelista V, Tacconelli S, Patrignani P. Effects of estrogen on endothelial prostanoid production and cyclooxygenase-2 and heme oxygenase-1 expression. Prostaglandins Other Lipid Mediat. 2012 Aug;98(3-4):122-8. doi: 10.1016/j.prostaglandins.2012.01.006. Epub 2012 Feb 6. PMID 22330859
- [Derived] Pauls SD, Du Y, Clair L, Winter T, Aukema HM, Taylor CG, Zahradka P. Impact of Age, Menopause, and Obesity on Oxylipins Linked to Vascular Health. Arterioscler Thromb Vasc Biol. 2021 Feb;41(2):883-897. doi: 10.1161/ATVBAHA.120.315133. Epub 2020 Dec 31. PMID 33380172
- [Derived] Gabbs M, Zahradka P, Taylor CG, Aukema HM. Time Course and Sex Effects of alpha-Linolenic Acid-Rich and DHA-Rich Supplements on Human Plasma Oxylipins: A Randomized Double-Blind Crossover Trial. J Nutr. 2021 Mar 11;151(3):513-522. doi: 10.1093/jn/nxaa294. PMID 33097936
- See also: Canadian Centre for Agri-Food Research in Health and Medicine — http://www.ccarm.ca